CLINICAL TRIAL: NCT04823585
Title: Aggravated Airway Inflammation: Research on Biological Treatment (Mepolizumab)
Acronym: AirGOs-biol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Salmi, Professor MD PhD Chief Physician, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUS/686/2020
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Asthma, Aspirin-Induced; Chronic Rhinosinusitis with Nasal Polyps
MeSH Terms: conditions — Asthma, Aspirin-Induced | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- subcutaneous injections of placebo (Placebo Comparator): Subcutaneous injections of placebo (physiological sodium chloride solution) once per month for 16 weeks. A total of 4 injections.
  Interventions: Drug: Placebo
- subcutaneous injections of Mepolizumab 100 mg (Experimental): Subcutaneous injections of Mepolizumab 100 mg once per month for 16 weeks. A total of 4 injections.
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — Solution. Subcutaneous. Mepolizumab is a biological drug, a humanized monoclonal antibody against interleukin-5.
  Arms: subcutaneous injections of Mepolizumab 100 mg
Drug: Placebo — Solution. Subcutaneous.
  Arms: subcutaneous injections of placebo

SUMMARY:
Primary objective:

to investigate the efficacy of Mepolizumab 100 milligram (mg) every month compared to placebo in reducing validated Sinonasal Outcome Test -22 score and on reducing endoscopic Nasal Polyp Score. The participants have a triad of chronic rhinosinusitis with nasal polyps (CRSwNP), asthma and non-steroidal anti-inflammatory drug exacerbated respiratory disease (NERD). The investigators will evaluate whether mepolizumab reduces the need for increased drug dosage (topical corticosteroid or bronchodilator dosage) and improves lung and nasal function more effectively than placebo.

This first visit ensures the inclusion and exclusion criteria of the subject. If necessary, NERD will be verified by an ASA challenge test at a second additional visit. Participants have also 6 visits, on four of which subcutaneous injection of the study product is administered. During visits, a clinical examination, airway function tests, and nasal, blood, urine, and stool samples are also taken to elucidate predictive biomarkers of severely symptomatic NERD patients.

DETAILED DESCRIPTION:
Primary objective:

to investigate the efficacy of Mepolizumab 100 milligram (mg) every month compared to placebo in reducing validated Sinonasal Outcome Test -22 score and on reducing endoscopic Nasal Polyp Score. The participants have a triad of chronic rhinosinusitis with nasal polyps (CRSwNP), asthma and non-steroidal anti-inflammatory drug exacerbated respiratory disease (NERD). The investigators will evaluate whether mepolizumab reduces the need for increased drug dosage (topical corticosteroid or bronchodilator dosage) and improves lung and nasal function more effectively than placebo.

This first visit ensures the inclusion and exclusion criteria of the subject. If necessary, NERD will be verified by an ASA challenge test at a second additional visit. Participants have also 6 visits, on four of which subcutaneous injection of the study product is administered. During visits, a clinical examination, airway function tests, and nasal, blood, urine, and stool samples are also taken to elucidate predictive biomarkers of severely symptomatic NERD patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Exacerbation of respiratory symptoms by acetylsalicylic acid (ASA) or another NSAID. (NERD will be verified by another visit if necessary).
* chronic rhinosinusitis with bilateral polyps. Endoscopic bilateral nasal polyp score of at least 5 (out of 8), with a minimum score of 2 in each nasal cavity
* Lund Mackay score ≥12 (maximum 24) of sinus computed tomography (CT) or cone beam (CBCT) scans. The new sinus CT/CBCT scans are needed if the previous sinus CT/CBCT scans have been performed over 36 months before recruitment visit or if there is a suspicion of complication of CRS (f.ex. mucocele, invasive fungal rhinosinusitis). Pregnant and breast-feeding subject will be excluded. Females of Reproductive Potential (FRPs) who are not pregnant or breast-feeding may be enrolled. FRPs need to perform pregnancy test prior to the CT/CBCT scans. If subject is already on contraception prior to the study this should be continued. The data of previous sinus CT/CBCT scans will be used if previous sinus CT/CBCT scans have been performed ≤36 months prior to recruitment visit. The clinical information of sinus CT/CBCT scans is critical to enrolling appropriate subjects for the research and cannot readily be obtained another way. The radiation dose of sinus CT/CBCT scans is less than 0.1 mSv, which corresponds to less than 10 days of natural background radiation in Finland. This dose has not been shown to increase the cancer risk.
* ≥1 previous CRS-surgery. Note that the last CRS-surgery must have been performed at least 6 months before 1st visit
* SNOT-22 ≥25
* At least one other symptom, such as partial loss of smell (hyposmia), nasal obstruction, total loss of smell (anosmia), or anterior or posterior rhinorrhea
* patient should have a history of at least one exacerbation during the past two years e.g. at least one criterion must be fulfilled of the following list during the past two years ≥1 oral corticosteroids; ≥3 antibiotic courses; ≥1 CRS-operation; ≥ 1 asthma hospitalization. In patients with contraindications of previously listed treatment or continuous oral steroids, additional criteria are not required.
* Asthma diagnosis (patient has the National Social Insurance Institution´s reimbursement right for asthma medication)
* Peripheral blood eosinophils (PBEos) >300 cells/ul at visit 1 OR (PBEos >150 cells/ul at visit 1 AND a history of PBEos >300 cells/ul during the past 12 months). A history of Nasal polyp tissue eosinophilia (NPeos) ≥30% during the past 12 months is a supportive criterion.

Exclusion Criteria:

* Age <18 years
* Age > 70 years
* CRS-surgery < 6 months before 1st visit
* pregnancy/ breastfeeding. FRPs need to perform pregnancy test prior to the CT/CBCT scans. If subject is already on contraception prior to the study this should be continued.
* complication of CRS (f.ex. mucocele, invasive fungal rhinosinusitis). Take sinus CT/CBCT scans, if needed!
* acute rhinosinusitis/respiratory infection
* severe disease related to airways/ immunology: cystic fibrosis, primary ciliary dyskinesia (PCD), sarcoidosis, immunosuppression, diagnosed Specific antibody deficiency (SAD), CVI, HIV, fungal rhinosinusitis; Young syndrome; Kartagener syndrome;
* other severe disease such as active cancer
* Received biologic therapy/systemic immunosuppressant/ASA desensitization therapy/experimental monoclonal antibody treatment to treat inflammatory or autoimmune disease within 2 months of study entry or 5 half-lives, whichever is longer. The patient is allowed to use ASA dose <100 mg/day due to cardiovascular reasons after ASA desensitization.
* current immunotherapy
* communication problems (f.ge. neurological/psychiatric disease, language skills)
* unlikely to comply
* ASA-challenge negative.
* History of hypersensitivity to mepolizumab or excipients in the formulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Change From Baseline at Week 16 in Sinonasal Outcome Test -22 (SNOT-22) Score | Baseline, Week 16
  SNOT-22 is a validated symptom questionnaire. The score ranges between 0 and 110. A higher score means worse outcome.
Change From Baseline at Week 16 in endoscopic Nasal polyp score of nasal cavity | Baseline, Week 16
  Nasal polyp score is graded based on polyp size from 0 = no polyps to 4 = large polyps causing complete obstruction of inferior nasal cavity. The score ranges between 0 and 110. A higher score means worse outcome.The Nasal polyp score FEV1% is measured by spirometry. A higher value means better lung function = better outcome.

SECONDARY OUTCOMES:
Change From Baseline at Week 16 in relative Forced expiatory volume in 1 second (FEV1 %) without bronchodilator. | Baseline, Week 16
  FEV1% is measured by spirometry. It is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration, in relation to the validated national reference value of subjects with similar age, gender and height.

CONTACTS AND LOCATIONS:
Overall Officials: Sanna Toppila-Salmi, MD PhD, PI, Principal Investigator — Helsinki University Hospital, Skin and Allergy Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Due to Finnish data protection legislation, confidential, health-related data, the datasets produced and/or examined during this study are not accessible to the general public. They can solely be managed by designated individuals within the study group for specific research objectives. The datasets analyzed during the current study are available from the corresponding author upon reasonable request. Data use permissions can be applied from the competent authorities.

REFERENCES:
- [Derived] Lyly A, Sahlman J, Pajala K, Salminen M, Sillanpaa S, Numminen J, Hanif T, Laulajainen-Hongisto A, Makela M, Kauppi P, Kangasniemi I, Lilja M, Hammaren-Malmi S, Virkkula P, Toppila-Salmi S. Study protocol for a randomized double-blinded placebo-controlled trial on mepolizumab for patients with chronic rhinosinusitis with nasal polyps, NSAID exacerbated respiratory disease and asthma. Front Allergy. 2025 Mar 21;6:1568081. doi: 10.3389/falgy.2025.1568081. eCollection 2025. PMID 40191526